CLINICAL TRIAL: NCT04956679
Title: Family-based Screening and Treatment of Helicobacter Pylori：A Real World Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of QiLu Hospital, Shandong University
Other Study IDs: 2019SDU-QILU-186
Record Dates: First submitted 2021-06-25; First posted 2021-07-09 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Helicobacter Pylori; Family
Keywords: Helicobacter pylori; Family

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family members in the study: Community groups that meet the inclusion criteria
  Interventions: Diagnostic Test: carbon 13 breath test

INTERVENTIONS:
Diagnostic Test: carbon 13 breath test — Patients with positive Helicobacter pylori infection were determined by carbon 13 breath test ,The diagnosis and treatment of positive patients were followed up without other intervention.

SUMMARY:
The habit of family meals makes the infection rate of Helicobacter pylori high in China, which is also the main cause of reinfection of Helicobacter pylori. Eating together can easily cause family members to be infected with Helicobacter pylori. We used a real-world study to understand the risk factors, epidemiological characteristics, and safety and effectiveness of eradication therapy for helicobacter pylori infection in family-based screening and treatment.

DETAILED DESCRIPTION:
Helicobacter pylori infection is a worldwide problem, which is the main cause of gastric cancer. The habit of sharing meals in the family is one of the factors contributing to the high infection rate of HP in China, as well as the main cause of reinfection of HP. Sharing meals can easily cause family members to be infected with HP.Family members live together, eat together, share tableware and other behaviors through the "mouth to mouth" transmission of Helicobacter pylori may be infected with each other, is also one of the reasons for the eradication of many patients after re-infection.At the same time, repeated infection and treatment of Helicobacter pylori will increase the difficulty of Helicobacter pylori reeradication.As a family unit, to study the status of our country family helicobacter pylori infection, epidemiological characteristics, infection risk factor, the different schemes, such as the safety and efficacy of treatment to take measures to reduce the infection rate is of great significance to prevention and treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Community population over 3 years old who signed the informed consent.
* at least 2 people in the family.
* living together for at least 10 months each year in the past 5 years except child aged below 5.

Exclusion Criteria:

* PPI drugs such as esomeprazole、pantoprazole、 rabeprazole,、lansoprazole、famotidine and H2 receptor antagonists were taken within two weeks.
* antibiotics、bismuth agents or traditional Chinese medicine with antibacterial effect were taken within four weeks
* There are other factors that researchers think are not suitable for participation

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community population aged above 3 years in family unit,The family unit is determined by actual living together rather than household registration relationship, with at least 2 people in the family and living together for at least 10 months each year in the past 5 years.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Patient compliance of performing medical examination. | 1 year
  Good compliance of medical examination advice was defined as the subjects took the medical advice given by the doctor and the rate of adoption and implementation of the medical examination advice.
Patient compliance of taking medication | 1 year
  Patient compliance of taking medication is defined as the ratio of the actual dose of medication taken by the patient to the total amount of medication required by the prescription. Good medication compliance is defined as the ratio greater than 80%.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 1 year
  Adverse reactions related to medication were recorded
Lesion detection ratio | 1 year
  The lesion detection ratio was defined as the ratio of the number of subjects who underwent medical examination on the basis of doctor's recommendation and were finally diagnosed with lesion to the number of subjects who underwent examination.
Eradication rate | 1 year
  Eradication rate was defined as the ratio of the number of patients diagnosed positive on the carbon 13 breath test to the number of subjects who turned negative after taking the eradication drug to the number of subjects diagnosed positive before taking the drug.

SECONDARY OUTCOMES:
The high-risk factors of Helicobacter pylori infection in families were investigated by questionnaire statistics. | 1 year
  Questionnaire survey was used to conduct information statistics on families undergoing Helicobacter pylori screening.Statistics include family members of the general situation, basic information, personal health and life habit, individual disease history, personal nearly 1 month medications, family health and lifestyle, family history, history of HP infection and the eradication of history, screening results, doctor give opinions and patient adherence and follow-up outcome after screening process, etc. Statistical soft ware was used to analyze factor correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,QiLu Hospital,Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546